CLINICAL TRIAL: NCT05162872
Title: A Phase II Study of Combination of Niraparib And Sintilimab In Recurrent/Metastatic Nasopharyngeal Carcinoma
Brief Title: Niraparib And Sintilimab In Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Professor of Medical Oncology, Director of Medical Oncology Department of Sun Yat-Sen University Cancer Centre (SYSUCC), Deputy Director of Lung Cancer Research Centre of SYSU, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-FXY-039
Record Dates: First submitted 2021-11-23; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PD-(L)1 naive patients, ≥1L of platinum-based chemotherapy (Experimental): Histologically confirmed recurrent or metastatic nasopharyngeal carcinoma (including recurrence and metastasis after radiotherapy, or a condition not suitable for surgery and radiotherapy judged by investigator)
  ≥ 1L of platinum-based chemotherapy at least 1 measurable lesion (RECIST 1.1) ECOG 0-1, PD-(L)1 naive patients, Niraparib 200 mg QD D1-21,Sintilimab 200 mg IV q3W, first step enroll N1=23 participants, if CR+PR≥3,then go to the second step, continue to enroll N2=39 participants, if CR+PR<3，then do not go to the second step.
  Interventions: Drug: Niraparib，Sintilimab
- PD-(L)1 previously treated patients，≥1L of platinum-based chemotherapy (Experimental): Histologically confirmed recurrent or metastatic nasopharyngeal carcinoma (including recurrence and metastasis after radiotherapy, or a condition not suitable for surgery and radiotherapy judged by investigator)
  ≥ 1L of platinum-based chemotherapy at least 1 measurable lesion (RECIST 1.1) ECOG 0-1, PD-(L)1 previously treated patients, Niraparib 200 mg QD D1-21,Sintilimab 200 mg IV q3W, first step enroll N1=20 participants, if CR+PR≥1,then go to the second step, continue to enroll N2=17 participants, if CR+PR<1，then do not go to the second step.
  Interventions: Drug: Niraparib，Sintilimab

INTERVENTIONS:
Drug: Niraparib，Sintilimab — Niraparib 200 mg QD D1-21 Sintilimab 200 mg IV q3W

SUMMARY:
this study is aimed to evaluate the efficacy and safety of the combination of Niraparib and Sintilimab in the treatment of recurrent/metastatic nasopharyngeal carcinoma

DETAILED DESCRIPTION:
this is a phase II, open-label study, to see whether the combination of Niraparib and Sintilimab is effective and safe to treat recurrent/metastatic nasopharyngeal carcinoma.

we will enroll patients who are histologically confirmed recurrent or metastatic nasopharyngeal carcinoma (including recurrence and metastasis after radiotherapy, or a condition not suitable for surgery and radiotherapy judged by investigator)

≥ 1L of platinum-based chemotherapy, at least 1 measurable lesion (RECIST 1.1), ECOG 0-1.

the study is designed to contain 2 cohorts: cohort A PD-(L)1 naive and cohort B PD-(L)1 previously treated patients, simon 2-steps design for each cohort, that is: for cohort A, first step will enroll 23 patients, if CR/PR patients ≥3， then go to the second step, continue to enroll 39 patients, otherwise this cohort ends. for cohort B, first step enroll 20 patients, if CR/PR patients ≥1，then continue to enroll 17 patients, otherwise the cohort ends.

Niraparib is a type of drug called a "PARP inhibitor", which blocks DNA (the genetic material of cells) damage from being repaired or may prevent damage from occurring in the first place. In cancer treatment, inhibiting PARP may help kill cancer cells by not allowing the cancer cells to repair its DNA damage or prevent DNA damage associated with nasopharyngeal carcinoma from occurring.

The FDA has not approved niraparib for nasopharyngeal carcinoma, but it has been approved for other uses.

ELIGIBILITY:
Inclusion Criteria:

* 1. A written informed consent form should be signed prior to any study-related procedures 2. Male or female, aged from 18~70 (inclusive) years 3. Histologically confirmed recurrent and/or metastatic nasopharyngeal carcinoma 4. At least 1 measurable lesion (RECIST 1.1 criteria) 5. Received ≥1L treatment (including but not limited to standard chemotherapy, targeted therapy, immunotherapy) ，with ≥1 platinum-based chemotherapy.

  6. ECOG score 0~1 7. Expected survival time ≥ 3 months 8. Good organ function includes:
* Neutrophil count≥1.5×109/L,
* Platelet count≥100×109/L,
* Hemoglobin≥9 g/dL
* Serum creatinine≤1.5×upper limit of normal (ULN), creatinine clearance≥60 mL/min (Cockcroft-Gault formula)
* Total bilirubin≤1.5×ULN
* AST and ALT≤2.5×ULN; for patients with liver metastasis, AST and ALT≤5×ULN, the investigator should determine whether they are enrolled
* Normal coagulation function: INR and PT≤1.5×ULN 9. Negative pregnancy test at enrollment. Male or female subjects should commit to take adequate and effective contraceptive measures or abstain from sexual for the duration of study participation and within 3 months after the last dose of the study drug 10. Toxicity of any previous chemotherapy have recovered to ≤ CTCAE Grade 1 or baseline 11. Other anti-tumor treatments have been discontinued, including but not limited to chemotherapy, radiotherapy, and surgery 4 weeks before receiving the study drug

Exclusion Criteria:

* 1. Known hypersensitivity to active or inactive ingredients of any drug in the study 2. Prior treatment with PARP inhibitors 3. Symptomatic and uncontrolled brain or leptomeningeal metastasis. No imaging scan is required to confirm no brain metastases 4. History of serious hypersensitivity reaction to any monoclonal antibody 5. Past or current diagnosis of MDS or AML 6. Major surgery within 4 weeks of starting the study or patient has not recovered from any effects of any major surgery 7. Patients with serious or uncontrolled diseases, including but not limited to:
* Uncontrollable nausea and vomiting, intestinal obstruction with symptoms that cannot be reduced, inability to swallow study drug, any gastrointestinal disorder that may interfere with drug absorption and metabolism
* Patients with respiratory syndrome due to pleural effusion or ascites (≥ CTCAE Grade 2 dyspnea)
* Active viral infections such as HIV, hepatitis B, hepatitis C, etc.
* Uncontrolled grand mal epilepsy, unstable spinal cord compression, superior vena cava syndrome, or other psychiatric disorders that affect the patient's signature of the informed consent form
* Immunodeficiency (other than splenectomy), or other condition that, in the opinion of the investigator, would expose the patient to high risk toxicity
* Active autoimmune disease or history of autoimmune disease that may recur and exert an effect on vital organ function or require treatment with immunosuppressive agents including systemic corticosteroids treatment period 8. Any systemic treatment requirement with corticosteroids (> 10 mg/day prednisone) or other immunosuppressive drugs within 14 days after receiving the study drug; in the absence of active autoimmune diseases, inhaled or topical steroids application and adrenal replacement doses (≤ 10 mg/day prednisone) are allowed; topical, intraocular, intra-articular, nasal, and inhaled corticosteroids (with small systemic absorption) are allowed; physiological replacement doses of systemic corticosteroids (≤ 10 mg/day prednisone) are allowed; the short-term corticosteroid therapy for the prevention (e.g., contrast allergy) or treatment of non-autoimmune diseases (e.g., delayed hypersensitivity caused by contact allergens) is allowed 9. History of bleeding tendency and thrombosis:
* Any bleeding event at CTCAE Grade 2 within 3 months prior to screening or at CTCAE Grade 3 or higher within 6 months prior to screening
* With active bleeding or coagulation abnormalities, bleeding tendency, or receiving thrombolytic or anticoagulation therapy
* Anticoagulation therapy is needed with warfarin or heparin
* Chronic antiplatelet therapy (e.g., aspirin, clopidogrel) is needed
* Thrombotic or embolic event within the past 6 months, e.g., cerebrovascular accident (including transient ischemic attack), and pulmonary embolism 10. Serious cardiovascular history:

  1. NYHA (New York Heart Association) Class 3 and 4 congestive heart failure
  2. Unstable angina or newly diagnosed angina or myocardial infarction within 12 months before screening
  3. Arrhythmia requiring therapeutic intervention (patients taking β-blockers or digoxin can be included)
  4. ≥ CTCAE Grade 2 valvular heart disease
  5. Hypertension that cannot be controlled with medication (systolic pressure > 150 mmHg or diastolic pressure > 100 mmHg) 11. Patients with any previous or current disease, treatment, or laboratory abnormality that may interfere with the results of the study and the throughout participation of the patient, or in the opinion of the investigator, the patient is not appropriate for the study; patients should not receive platelet or red blood cell infusions 4 weeks before the start of treatment with study drug 12. Patients who are pregnant or lactating, or who intend to become pregnant during the study treatment period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 180 days.
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR).

SECONDARY OUTCOMES:
DoR | up to 180 days.
  DoR was defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of disease progression or to death due to any cause, whichever occurred first.
DCR | up to 180 days.
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) and Stable Disease(SD).
PFS | up to 180 days.
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
OS | up to 360 days.
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Li zhang, DOCTOR, Principal Investigator — SUN YAT-SEN UNVERISITY CANCER CENTER
Locations (1):
- Li zhang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No